CLINICAL TRIAL: NCT00005776
Title: The Randomized Inhaled Nitric Oxide Study (NINOS) in Full-Term and Nearly Full-Term Infants With Hypoxic Respiratory Failure
Brief Title: Inhaled Nitric Oxide Study for Respiratory Failure in Newborns
Acronym: NINOS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Results showed statistically significant benefit in the experimental group
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Medical Research Council of Canada (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Richard A. Ehrenkranz, NRN Lead Study Investigator, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0014; U01HD019897 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD021415 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027881 (NIH); U10HD027904 (NIH); U10HD034167 (NIH); U10HD034216 (NIH); M01RR000070 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR001032 (NIH); M01RR006022 (NIH); M01RR008084 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome; Pneumonia, Aspiration; Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency
Keywords: NICHD Neonatal Research Network; Hypertension, pulmonary; Hypoxic respiratory failure; Meconium aspiration; Methemoglobinemia; Nitric oxide; Oxygen inhalation therapy; Persistent Fetal Circulation Syndrome; Pneumonia, aspiration; Respiratory distress syndrome; Respiratory insufficiency; Severe respiratory failure
MeSH Terms: conditions — Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome; Pneumonia, Aspiration; Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency; Meconium Aspiration Syndrome; Methemoglobinemia; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled Nitric Oxide (iNO)
  Interventions: Drug: Inhaled nitric oxide
- Oxygen (Placebo Comparator): 100% oxygen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled nitric oxide — Inhaled Nitric oxide at a concentration of 20 ppm
  Arms: Inhaled Nitric Oxide
Drug: Placebo — 100% Oxygen
  Arms: Oxygen

SUMMARY:
Respiratory failure in term newborns is associated with increased rates of death and long-term neurodevelopmental problems. This large international multicenter trial randomized newborns who had failed to respond to intensive care, including high levels of ventilator support, to receive either inhaled nitric oxide (iNO) or 100 percent oxygen to test whether iNO would decrease their risk of dying or requiring temporary lung bypass. Infants were followed during their initial hospitalization; their outcome was assessed at 18 to 24 mos of age.

DETAILED DESCRIPTION:
Respiratory failure in term newborns is associated with significant morbidity and mortality, despite maximal conventional therapy. Neonates with pulmonary hypertension have been treated with iNO, a selective pulmonary vasodilator. This multicenter, double-masked placebo-controlled randomized trial tested whether iNO would reduce the risk of death and/or the initiation of extracorporeal membrane oxygenation (ECMO) in a prospectively defined cohort of term or near-term neonates with hypoxic respiratory failure unresponsive to conventional therapy. The sample size was based on a reduction of the primary event (death or ECMO) from 50 percent to 30 percent; 90 percent power; and a two-tailed Type I error of 0.05.

Infants were evaluated at baseline for pulmonary, cardiac, bleeding status, and therapies received. Those who were greater than 34 wks gestation and 14 days old or less and required assisted ventilation with an OI (mean airway pressure x FiO2 divided by the PaO2 x 100) greater than 25 were eligible. They were randomly assigned to receive iNO at 20 ppm or 100 percent oxygen as a control. Infants whose PaO2 increased by less than 20 mm Hg after 30 minutes were studied at 80ppm iNO or control gas.; MetHg and NO2 concentrations were monitored regularly. Management, including surfactant administration, included prospectively defined criteria for study gas response, escalation, reinitiation, and weaning. The maximum total time on study gas was 336 hrs (after 240 hrs, the INO concentration was required to be no more than 5 ppm). Patients were followed to death, discharge, or 120 days and evaluated at 18-24 mos by a masked certified examiner.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 34 wks gestational age
* One or more of the following diagnoses: primary pulmonary hypertension of the newborn, respiratory distress syndrome, perinatal aspiration syndrome, pneumonia/sepsis, suspected pulmonary hypoplasia
* Oxygenation Index (OI) greater than 15 and less than 25 on 2 arterial blood gases at least 15 min apart
* Indwelling arterial line
* Echocardiography before randomization
* Parental consent

Exclusion Criteria:

* Congenital diaphragmatic hernia
* Known congenital heart disease
* Decision not to provide full therapy

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 1995-10; Primary Completion 1996-05 (Actual); Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Death or initiation of ECMO | Before hospital discharge or 120 days of life

SECONDARY OUTCOMES:
PaO2 levels, oxygenation index, and alveolar-arterial oxygen gradient | 30 minutes after drug administration
Neurodevelopmental outcome | 18-22 Months Corrected Age
Duration of hospital stay | At hospital discharge
Duration of assisted ventilation, air leaks, or chronic lung disease | At hospital discharge
Transfers for ECMO | At hospital discharge
Meeting ECMO criteria | At hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Ehrenkranz, MD, Study Director — Yale University; David K. Stevenson, MD, Principal Investigator — Stanford University; Raymond Bain, PhD, Principal Investigator — George Washington University; James A. Lemons, MD, Principal Investigator — Indiana University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; William William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Mary Wearden, MD, Principal Investigator — Baylor College of Medicine; N. Singhal, MD, Principal Investigator — Foothills Hospital, Calgary, Canada; Neil N. Finer, MD, Principal Investigator — Royal Alexandra Hospital; A. Solimano, MD, Principal Investigator — British Columbia Children's Hospital; C. Fajardo, MD, Principal Investigator — Health Sciences Center, Winnipeg, Manitoba; H. Kirpalani, MD, Principal Investigator — McMaster University; R. Walker, MD, Principal Investigator — Children's Hospital of Eastern Ontario; A. Johnston, MD, Principal Investigator — Montreal Children's Hospital of the MUHC; P. Blanchard, MD, Principal Investigator — Université de Sherbrooke, Sherbrooke, Quebec; K. Sankarhan, MD, Principal Investigator — Royal University Hospital, Saskatoon, Saskatchewan
Locations (20):
- United States (11):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
- Canada (9):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Université de Sherbrooke,, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Neonatal Inhaled Nitric Oxide Study Group. Inhaled nitric oxide in full-term and nearly full-term infants with hypoxic respiratory failure. N Engl J Med. 1997 Feb 27;336(9):597-604. doi: 10.1056/NEJM199702273360901. PMID 9036320
- [Result] Inhaled nitric oxide and hypoxic respiratory failure in infants with congenital diaphragmatic hernia. The Neonatal Inhaled Nitric Oxide Study Group (NINOS). Pediatrics. 1997 Jun;99(6):838-45. doi: 10.1542/peds.99.6.838. PMID 9190553
- [Result] Inhaled nitric oxide in term and near-term infants: neurodevelopmental follow-up of the neonatal inhaled nitric oxide study group (NINOS). J Pediatr. 2000 May;136(5):611-7. doi: 10.1067/mpd.2000.104826. PMID 10802492
- [Result] Sokol GM, Fineberg NS, Wright LL, Ehrenkranz RA. Changes in arterial oxygen tension when weaning neonates from inhaled nitric oxide. Pediatr Pulmonol. 2001 Jul;32(1):14-9. doi: 10.1002/ppul.1083. PMID 11416871
- [Result] Sokol GM, Ehrenkranz RA. Inhaled nitric oxide therapy in neonatal hypoxic respiratory failure: insights beyond primary outcomes. Semin Perinatol. 2003 Aug;27(4):311-9. doi: 10.1016/s0146-0005(03)00043-0. PMID 14510322
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org